CLINICAL TRIAL: NCT02393508
Title: The Impact of Red Cell Age on Product Utilization in the Chronically Transfused Outpatient Population
Acronym: ABC-TOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oksana Prokopchuk-Gauk, Transfusion Medicine Fellow (Co-Investigator), University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-16748
Record Dates: First submitted 2015-03-05; First posted 2015-03-19 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Bone Marrow Failure Syndrome
Keywords: transfusion, red blood cell; transfusion reaction; quality of life
MeSH Terms: conditions — Bone Marrow Failure Disorders; Transfusion Reaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh Human Red Blood Cells (Active Comparator): Participants will receive transfusion of human donor red blood cells that are less than or equal to 7 days of age from the time of donation.
  Interventions: Other: Fresh Human Red Blood Cells
- Aged Human Red Blood Cells (Active Comparator): Participants will receive transfusion of human donor red blood cells that are greater than 21 days and up to a maximum of 42 days of age from the time of donation.
  Interventions: Other: Aged Human Red Blood Cells

INTERVENTIONS:
Other: Fresh Human Red Blood Cells — Red cell units for transfusion will be acquired from Canadian Blood Services (CBS), as a part of their usual stock to the Calgary Zone. Blood will be processed and prepared by CBS according to their standard protocol. The red cell units assigned to patients as a part of this trial will not be manipulated in any way prior to participant transfusion.
  Arms: Fresh Human Red Blood Cells
Other: Aged Human Red Blood Cells — Red cell units for transfusion will be acquired from Canadian Blood Services (CBS), as a part of their usual stock to the Calgary Zone. Blood will be processed and prepared by CBS according to their standard protocol. The red cell units assigned to patients as a part of this trial will not be manipulated in any way prior to participant transfusion.
  Arms: Aged Human Red Blood Cells

SUMMARY:
In this study, the investigators will be evaluating the impact of red blood cell age in patients receiving chronic blood transfusions in the outpatient setting. This study will have a double-bind, randomized trial design, meaning that the investigators and participants will not be told the group assignment at study enrollment.

Study participants will be randomly divided into two groups (50% of participants in each group) by a computer generated block randomization schema. The 'fresh blood' group will receive blood units that are 7 or less from the time of donor collection, and the 'aged blood' group will receive blood units that are greater than 21 to 42 days from the time of donor collection. The number of units of blood transfused will be decided based on the participant's hemoglobin level before blood transfusion.

The primary goal of our study is to compare annual red blood cell product use (the number of units given per patient in a year). The investigators will also be comparing groups to evaluate the transfusion reaction frequency, iron burden (based on the level of ferritin in the blood), overall transfusion and care cost difference, and participant time spent in outpatient departments.

Our hypothesis is that use of fresh blood in chronically transfused patients will lead to a decrease the in red cell transfusion rate, with subsequent clinical benefits including reduction of transfusion reaction frequency and systemic iron burden.

This study will be taking place within the Calgary Zone of Alberta Health Services only.

DETAILED DESCRIPTION:
Background: Chronically transfused medical outpatients comprise a significant proportion of transfusion recipients annually. At this time, the impact of red cell transfusion on patient outcomes in this patient population is unknown.

Objective: Our goal is to prospectively evaluate impact of red cell age on product utilization in a cohort of chronically transfused medical outpatients randomized to receive red blood cells that are fresh (≤ 7 days from collection) or aged (>21-42 days from collection). To our knowledge, no other studies with a similar design or objective have been published.

Patient population and study design: Patients meeting eligibility criteria will be invited to participate in our study. Our chronically transfused outpatient population is defined as adults who are receiving 2 or more red cell units per month for at least 3 consecutive months in an ambulatory clinic setting within the Calgary Zone.

We plan to incorporate both prospective and retrospective data collection and analysis in our study design. All eligible, consenting participants will be randomized into one of the two study arms. Investigators and participants will be blinded to participant group assignment.

Laboratory parameters and red cell transfusion: Parameters of usual pre-transfusion bloodwork will be followed, including complete blood count (CBC) and ferritin levels. Red cell transfusion volumes for chronic transfusion throughout the study will be determined according to a locally established protocol to achieve a post-transfusion hemoglobin (Hb) of 95-105 g/dL. Given that 1 adult unit of red cells raises the baseline Hb by approximately 10 g/L, the following volumes will be given to patients during a single visit based on their pre-transfusion CBC: Hb <75 = 3 units, Hb 75-84 = 2 units, Hb 85-94 = 1 unit, Hb ≥95 = no transfusion. A routine post-transfusion CBC will not be performed. According to usual care, participants will have a standing order to perform a CBC at least weekly, or if they have subjective symptoms of anemia to help guide subsequent transfusions.

Study participants will receive blood transfusion in usual locations designated within the Calgary Zone for administration of chronic blood transfusions. These include medical daycare units at the Foothills Medical Center, Tom Baker Cancer Center, Peter Lougheed Center, and South Health Campus. Nurses will administer blood transfusions according to standard practice, without change in transfusion protocol despite patient study participation.

Duration of participation will be 1 year from the time of enrollment. Participant health record access will be required for collection of demographic information and retrospective data involving any transfusions received within 1 year prior to enrollment to establish transfusion chronicity and health patterns. Outcomes will be based on a comparison of results between the study groups. Prospectively collected data based on red cell age will additionally be compared to retrospective transfusion related information (including red cell transfusion frequency and blood age) from within 1 year from the time of enrollment, if available. We plan to enroll a maximum total of 60 participants, with assignment of 30 patients into each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring outpatient chronic red cell transfusions (2 or more red blood cell units per month for at least 3 consecutive months) in an ambulatory clinic within the Calgary Zone

Exclusion Criteria:

* prerequisite for fresh or irradiated blood due to a pre-existing medical reason
* hemodialysis dependence
* chronic disease that has acutely decompensated, with a life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Red blood cell transfusion rate | 1 year from the time of enrollment
  Product utilization, comparing the number and frequency of red blood cell units transfused to the chronically transfused outpatient population eligible for trial participation

SECONDARY OUTCOMES:
Ferritin burden | At enrollment, 3 months, 6 months, 9 months and 12 months
  Based on results of laboratory test results available in the participant's electronic medical record, as ordered as a part of standard care by the primary hematologist
Total cost of blood product transfusion | 1 year from the time of enrollment
  Approximate sum of the cost of blood products transfused and nursing services required in the outpatient hospital treatment rooms when transfusions are administered throughout the study period
Number of hours spent receiving blood products | 1 year from the time of enrollment
  Sum of the number of patient hours spent receiving transfusions in the hospital treatment room setting
Transfusion reaction frequency | 1 year from the time of enrollment
  Number and type of transfusion reactions experienced by patients receiving transfusions throughout the study period, as reported to transfusion medicine by nursing, according to standard practice protocols

CONTACTS AND LOCATIONS:
Overall Officials: Meer-Taher Shabani-Rad, MD, FRCPC, Principal Investigator — University of Calgary

REFERENCES:
- [Background] Hebert PC, Chin-Yee I, Fergusson D, Blajchman M, Martineau R, Clinch J, Olberg B; Canadian Critical Care Trials Group. A pilot trial evaluating the clinical effects of prolonged storage of red cells. Anesth Analg. 2005 May;100(5):1433-1458. doi: 10.1213/01.ANE.0000148690.48803.27. PMID 15845701
- [Background] Taylor RW, O'Brien J, Trottier SJ, Manganaro L, Cytron M, Lesko MF, Arnzen K, Cappadoro C, Fu M, Plisco MS, Sadaka FG, Veremakis C. Red blood cell transfusions and nosocomial infections in critically ill patients. Crit Care Med. 2006 Sep;34(9):2302-8; quiz 2309. doi: 10.1097/01.CCM.0000234034.51040.7F. PMID 16849995
- [Background] Weinberg JA, McGwin G Jr, Griffin RL, Huynh VQ, Cherry SA 3rd, Marques MB, Reiff DA, Kerby JD, Rue LW 3rd. Age of transfused blood: an independent predictor of mortality despite universal leukoreduction. J Trauma. 2008 Aug;65(2):279-82; discussion 282-4. doi: 10.1097/TA.0b013e31817c9687. PMID 18695462
- [Background] Spinella PC, Carroll CL, Staff I, Gross R, Mc Quay J, Keibel L, Wade CE, Holcomb JB. Duration of red blood cell storage is associated with increased incidence of deep vein thrombosis and in hospital mortality in patients with traumatic injuries. Crit Care. 2009;13(5):R151. doi: 10.1186/cc8050. Epub 2009 Sep 22. PMID 19772604
- [Background] Koch CG, Li L, Sessler DI, Figueroa P, Hoeltge GA, Mihaljevic T, Blackstone EH. Duration of red-cell storage and complications after cardiac surgery. N Engl J Med. 2008 Mar 20;358(12):1229-39. doi: 10.1056/NEJMoa070403. PMID 18354101
- [Background] Mynster T, Nielsen HJ. The impact of storage time of transfused blood on postoperative infectious complications in rectal cancer surgery. Danish RANX05 Colorectal Cancer Study Group. Scand J Gastroenterol. 2000 Feb;35(2):212-7. doi: 10.1080/003655200750024416. PMID 10720122
- [Background] Yuruk K, Milstein DM, Bezemer R, Bartels SA, Biemond BJ, Ince C. Transfusion of banked red blood cells and the effects on hemorrheology and microvascular hemodynamics in anemic hematology outpatients. Transfusion. 2013 Jun;53(6):1346-52. doi: 10.1111/j.1537-2995.2012.03905.x. Epub 2012 Sep 24. PMID 22998160
- [Background] Triulzi DJ, Yazer MH. Clinical studies of the effect of blood storage on patient outcomes. Transfus Apher Sci. 2010 Aug;43(1):95-106. doi: 10.1016/j.transci.2010.05.013. Epub 2010 Jul 24. PMID 20656558